CLINICAL TRIAL: NCT00026104
Title: A Randomized Phase II Trial of Weekly Gemcitabine, Paclitaxel and External Irradiation (50.4 GY) Followed by the Farnesyl Transferase Inhibitor R115777 (NSC #702818) for Locally Advanced Pancreatic Cancer
Brief Title: Combination Chemotherapy Plus Radiation Therapy With or Without Tipifarnib in Treating Patients With Locally Advanced Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02423; RTOG-PA-0020; CDR0000068986; U10CA021661 (NIH)
Record Dates: First submitted 2001-11-09; First posted 2003-01-27 (Estimated); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Adenocarcinoma of the Pancreas; Stage II Pancreatic Cancer; Stage III Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Paclitaxel; Taxes; tipifarnib; Radiotherapy; Radiation

ARMS (2):
- Arm I (radiation therapy, paclitaxel, gemcitabine) (Experimental): Patients receive radiotherapy once daily, 5 days a week, for 5.5 weeks, beginning on day 1. Patients also receive paclitaxel IV over 1 hour and gemcitabine IV over 30 minutes on days 1, 8, 15, 22, 29, and 36.
  Interventions: Drug: gemcitabine hydrochloride; Drug: paclitaxel; Radiation: radiation therapy
- Arm II (radiation therapy, tipifarnib) (Experimental): Patients receive chemoradiotherapy as in arm I. Within 3-8 weeks after completion of chemoradiotherapy, patients without disease progression receive oral tipifarnib twice daily for 21 days.
  Interventions: Drug: tipifarnib; Radiation: radiation therapy

INTERVENTIONS:
Drug: gemcitabine hydrochloride — Given IV
  Other Names: dFdC; difluorodeoxycytidine hydrochloride; gemcitabine; Gemzar
  Arms: Arm I (radiation therapy, paclitaxel, gemcitabine)
Drug: paclitaxel — Given IV
  Other Names: Anzatax; Asotax; TAX; Taxol
  Arms: Arm I (radiation therapy, paclitaxel, gemcitabine)
Drug: tipifarnib — Given orally
  Other Names: R115777; Zarnestra
  Arms: Arm II (radiation therapy, tipifarnib)
Radiation: radiation therapy — Undergo radiation therapy
  Other Names: irradiation; radiotherapy; therapy, radiation

SUMMARY:
Randomized phase II trial to compare the effectiveness of gemcitabine, paclitaxel, and radiation therapy with or without tipifarnib in treating patients who have locally advanced pancreatic cancer. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Tipifarnib may stop the growth of tumor cells by blocking the enzymes necessary for tumor cell growth. Combining chemotherapy and radiation therapy with tipifarnib may be an effective treatment for pancreatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Compare the 1-year survival rate in patients with locally advanced pancreatic cancer treated with paclitaxel, gemcitabine, and radiotherapy with or without tipifarnib.

II. Determine the toxicity and loco-regional activity of this chemoradiotherapy regimen in these patients.

III. Determine the feasibility and toxicity of prolonged administration of tipifarnib after chemoradiotherapy in these patients.

IV. Determine whether tipifarnib administered after chemoradiotherapy can increase progression-free and overall survival in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to weight loss in the preceding 6 months (more than 10% vs 10% or less) and tumor dimension (at least 5 cm vs less than 5 cm). Patients are randomized to 1 of 2 treatment arms.

Arm I: Patients receive radiotherapy once daily, 5 days a week, for 5.5 weeks, beginning on day 1. Patients also receive paclitaxel IV over 1 hour and gemcitabine IV over 30 minutes on days 1, 8, 15, 22, 29, and 36.

Arm II: Patients receive chemoradiotherapy as in arm I. Within 3-8 weeks after completion of chemoradiotherapy, patients without disease progression receive oral tipifarnib twice daily for 21 days.

Treatment continues every 28 days in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed unresectable, locally advanced adenocarcinoma of the pancreas

  * Residual disease after resection (R1 or R2, microscopic or macroscopic) allowed
* No metastases in major viscera
* No peritoneal seeding or ascites
* Biliary or gastroduodenal obstruction must have drainage before starting study therapy
* Radiographically assessable disease encompassable within a single irradiation field (15 by 15 cm maximum)
* Performance status - Zubrod 0-1
* Granulocyte count at least 1,800/mm^3
* Platelet count at least 100,000/mm^3
* ALT less than 3 times upper limit of normal
* Bilirubin less than 2.0 mg/dL
* Creatinine less than 3.0 mg/dL
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other malignancy within the past 2 years except non-melanoma skin cancer or carcinoma in situ of the cervix, uterus, or bladder
* No significant infection or other medical condition that would preclude study
* No prior chemotherapy (including gemcitabine or paclitaxel) for pancreatic cancer
* No other concurrent cytotoxic agents
* See Disease Characteristics
* No prior radiotherapy to the planned field
* No other concurrent radiotherapy
* See Disease Characteristics
* No other concurrent investigational agents

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2001-11; Primary Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Overall survival | 1 year
  Calculated along with associated 95% confidence intervals.

SECONDARY OUTCOMES:
Frequency of patients developing unacceptable toxicity defined as grade 3 or higher gastrointestinal or pulmonary toxicity and/or discontinuation of treatment | Up to 5 years
  Graded according to the CTCAE version 3.0.
Difference in overall survival between treatment regimens | 1 year
  Estimated with a 95% confidence interval.
Progression-free survival | 1 year
  Calculated along with associated 95% confidence intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Tyvin Rich, Principal Investigator — Radiation Therapy Oncology Group
Locations (1):
- Radiation Therapy Oncology Group, Philadelphia, Pennsylvania, United States